CLINICAL TRIAL: NCT06055751
Title: Long Term Evaluation of Cardiac Arrhythmias After Transcatheter Aortic Valve Implantation -The LOCATE Registry
Status: Recruiting | Type: Observational
Sponsor: Kansas City Heart Rhythm Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: KCHRRF-LUX TAVR-0019
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Aortic Stenosis; Atrial Fibrillation New Onset; Heart Block
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Transcatheter aortic valve replacement (TAVR) with Boston Scientific Loop Recorder: This is a group of patients who have undergone TAVI procedure and implantation of Boston Scientific Loop Recorder (LUX-Dx PMA# K193473).
  Interventions: Device: TAVR Procedure and implantation of Boston Scientific Loop Recorder (LUX-Dx PMA# K193473)

INTERVENTIONS:
Device: TAVR Procedure and implantation of Boston Scientific Loop Recorder (LUX-Dx PMA# K193473) — No intervention will be done as part of this prospective registry. Implantation of Boston Scientific Loop Recorder (LUX-Dx) will be performed regardless of this research and outside this research protocol per standard of care

SUMMARY:
The purpose of the Long term Evaluation of Cardiac Arrhythmias after Transcatheter Aortic Valve Implantation (LOCATE) Registry is to perform long-term ambulatory monitoring of patients with severe aortic stenosis who undergo trans-catheter aortic valve implantation (TAVI) and develop new onset conduction system abnormalities post-procedure that do not require urgent permanent pacemaker (PPM) implantation. The primary objectives of this study are to assess the incidence of late onset heart block necessitating PPM implantation and to evaluate the incidence of new onset atrial fibrillation (AF) following TAVI. This study aims to provide valuable insights into the long-term cardiac health of TAVI patients and inform the development of improved treatment strategies for aortic stenosis patients with conduction system abnormalities.

DETAILED DESCRIPTION:
Clinical management of the patients that develop conduction system abnormalities not severe enough to warrant a PPM implantation is uncertain due to limited prospective long-term data on outcomes in this patient population with significant variations in treatment approaches. While some electrophysiologists favor ambulatory monitoring with event monitors or Implantable loop recorder (ILR), small studies have shown a potential benefit of invasive electrophysiological studies for risk stratification. Most rhythm monitoring studies have only focused on arrhythmias in the first 2-4 weeks post implantation with very sparse data on longer term outcomes. In addition to conduction system abnormalities, other arrhythmias such as AF following TAVI have also been shown to be associated with worse long-term outcomes. However, prospective data on incidence and risk factors of post TAVI atrial fibrillation is limited.

This will be a prospective observational study (Registry). Patients that have undergone a TAVI procedure and meet inclusion and no exclusion criteria will be approached about participating in the study. Patients who have undergone Boston Scientific Loop Recorder (LUX-Dx Premarket Approval Application (PMA)# K193473) as standard of care for arrhythmia monitoring after TAVI will have the ILR monitored monthly by the electrophysiology team. All alerts will be reviewed and discussed with the implanting physician for further management. Patients will be followed for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age with severe aortic stenosis that undergo TAVI for severe aortic stenosis that develop any one of the following conduction system abnormalities on the immediate post procedural or post operative ECG and have undergone ILR implantation for long-term monitoring of these conditions:
* New left bundle branch block (QRS >120ms)
* New first degree AV block (PR>200ms) or worsening of pre-existing first-degree AV block by >30ms
* New right bundle branch block (QRS>120ms)
* Intra-procedural 2:1 or higher-grade AV block with spontaneous improvement within 24 hours

Exclusion Criteria:

* Patients with high grade or complete AV block post TAVI needing urgent pacemakers
* Patient with existing cardiac implantable electronic devices (CIEDs)
* Patients having a particular medical condition that dictates that they cannot tolerate subcutaneous, chronically-inserted device
* Patient is currently pregnant as evidenced by urine positive Beta-HCG. (Urine Beta human chorionic gonadotropin (HCG) will be checked in all females of the reproductive age group).
* Patients not willing to sign the consent, lacks the capacity to sign the consent or revoke the consent after signing will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone Boston Scientific Loop Recorder (LUX-Dx PMA# K193473) as standard of care for arrhyhtmia monitoring after TAVI procedure will have the ILR monitored monthly by the electrophysiology team. All alerts will be reviewed and discussed with the implanting physician for further management. Patients will be followed for up to 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of brady arrhythmias | 12 Months
  Incidence of significant brady arrhythmias (2:1 or higher-grade Atrioventricular block (AV) block) requiring pacemaker implantation post TAVI in patients with evidence of conduction system injury following TAVI
Predictors of development of late onset heart block needing pacing | 12 Months
  Evaluate predictors of development of late onset (>30 days) heart block needing pacing
New onset Atrial Fibrillation | 12 Months
  Assess the incidence of new onset atrial fibrillation post TAVI

CONTACTS AND LOCATIONS:
Overall Officials: Naga Venkata K. Pothineni, MD, Principal Investigator — Kansas City Heart Rhythm Institute
Locations (2):
- United States (2):
  - Research Medical Center Clinic, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri

REFERENCES:
- [Background] Massoullie G, Ploux S, Souteyrand G, Mondoly P, Pereira B, Amabile N, Jean F, Irles D, Mansourati J, Combaret N, Mechulan A, Badoz M, Da Costa A, Defaye P, Motreff P, Clerfond G, Bordachar P, Eschalier R. Incidence and management of atrioventricular conduction disorders in new-onset left bundle branch block after TAVI: A prospective multicenter study. Heart Rhythm. 2023 May;20(5):699-706. doi: 10.1016/j.hrthm.2023.01.013. Epub 2023 Jan 13. PMID 36646235
- [Background] Lilly SM, Deshmukh AJ, Epstein AE, Ricciardi MJ, Shreenivas S, Velagapudi P, Wyman JF. 2020 ACC Expert Consensus Decision Pathway on Management of Conduction Disturbances in Patients Undergoing Transcatheter Aortic Valve Replacement: A Report of the American College of Cardiology Solution Set Oversight Committee. J Am Coll Cardiol. 2020 Nov 17;76(20):2391-2411. doi: 10.1016/j.jacc.2020.08.050. Epub 2020 Oct 21. PMID 33190683